CLINICAL TRIAL: NCT04620720
Title: Post Operative Pain in Modified Radical Mastectomy.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Anum Arif, Dr Anum Arif, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DUHSKK
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): routuine analgesics wil be given
- intervention group (Experimental): patient will receive cap gabapentin 1200 mg 2 hours before surgery
  Interventions: Drug: capule gabapentin

INTERVENTIONS:
Drug: capule gabapentin — neuropathic analgesic
  Arms: intervention group

SUMMARY:
we will assess post operative pain after surgery of modified radical mastectomy at 12 and 24 hours post operatively on arm movement and on rest

DETAILED DESCRIPTION:
This Randomised control trial will be conducted at the Department of General Surgery, Dow University Hospital OJHA Campus Karachi over a period of a year. All Females, ages ranged between 20 to 80 years and diagnosed with breast carcinoma stage II on the basis of triple assessment will be recruited in the study. Patients who will refuse to participate in the study, allergic to gabapentin on the basis if history, previous treatment with Gabapentin in the previous 8 weeks, Chronic pain syndrome, Substance abuse, sedatives, hypnotics or antidepressants, analgesic intake within 48 hours before surgery, Diabetes mellitus, Hypertension, and Acute or Chronic Renal Failure on the basis of medical records and Inability to understand VAS pain score will be excluded from the study. The sample size will be calculated by the Open Epi calculator. The mean pain score difference at rest between two groups was taken as 0.7 (Placebo: mean ± SD = 2.9 ± 1.2 and Gabapentin: mean ± SD = 2.2 ± 1.3.5 With 80% power, and 95% confidence level, the total sample size came out to be 102, 51 patients in each group. Consecutive sampling was used to achieve the desired sample. Patients fulfilling inclusion criteria were randomly enrolled in either of the 2 groups by sealed opaque envelop method bearing cards, which will be picked by the staff nurses. The intervention group was labeled as group A and the control group as group B. Patients in the intervention group received a single dose of 1200 mg of gabapentin 2hours before surgery. All procedures were performed under general anesthesia. Postoperative analgesic injection ketorolac 30 mg thrice a day and injection paracetamol 1 gram intravenous thrice a day was advised. Patients were assessed at 12 and 24 h post-operatively for pain scores at rest and arm mobilization using VAS pain score, a number of times rescue analgesia when VAS score > 3 by residents of surgery blinded to the study. Those patients, who experience pain (pain score > 3) in spite of routine analgesics received injection ketorolac 30 mg once, pain score between 3 to 6 received injection Kinz, pain score > 7 will be given both analgesics single times, pain score >8 will receive intravenous maximum thrice in 24 hours. Patients with pain score 0-2 will not be given any additional analgesic All patients will receive antiemetic in Metoclopramide 10 mg I.V in case of nausea and vomiting. All demographics and outcome variables will be entered in the proforma. The outcome variables of the study were age, pain score (VAS), and analgesic requirement.

ELIGIBILITY:
Inclusion Criteria:

* All Females, age ranged between 20 to 80 years and diagnosed with breast carcinoma stage II on the basis of triple assessment will be recruited in the study

Exclusion Criteria:

* Patients who will refuse to participate in the study, allergic to gabapentin on the basis if history, previous treatment with Gabapentin in previous 8 weeks , Chronic pain syndrome, Substance abuse, sedatives, hypnotics or antidepressants ,analgesic intake within 48 hours before surgery, Diabetes mellitus, Hypertension and Acute or Chronic Renal Failure on the basis of medical records

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain score | 12 hours post oepratively
  Visual analog score for pain from 0 to 10. O means no pain. 1 is least and 10 is most severe pain

SECONDARY OUTCOMES:
analgesia requirement | 12 hours post oepratively
  change in analgesic requirement a i either groups

CONTACTS AND LOCATIONS:
Overall Officials: Anum Arif, MBBS FCPS, Principal Investigator — Combined military hospital lahore
Locations (1):
- Anum, Karachi, Select A State Or Province, Pakistan

IPD SHARING:
Plan to Share IPD: No